CLINICAL TRIAL: NCT07354360
Title: Effect of Oketani Massage on Successful Breastfeeding
Brief Title: Effect of Oketani Breast Massage on Promoting Breastfeeding
Acronym: OKETANI-BF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NURS-MU-OKETANI-2026
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Breastfeeding; Massage; Breastfeeding Self-Efficacy; Oketani Massage
Keywords: Breastfeeding; Oketani massage; breastfeeding self-efficacy; breast engorgement; Feeding Behavior
MeSH Terms: conditions — Breast Feeding; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: * The massage will be performed very gently and rhythmically on the right and left breasts within 8 several manual steps. From one to seven refers to (the course of treatment) & Step eight refers to (milking or expressing).
  * One minute will be spent on a series of tasks and statements, which will be repeated for 15 to 20 minutes. Pushing and pulling away included manipulations in stages one, two, and three will be carried out gently and painlessly on primipara women in order to separate the hard section of the breast from the fascia of the pectoralis. Four to six steps will be required to drag the entire breast downward and to either side with two thumbs and two hands. At four Steps; the total breast will be pushed down towards the umbilicus. Five to six steps will be done to disconnect the hard base parts of the breast. In addition to, the breast will be circulated clockwise in the first seven steps with an expansion of its base. In the eighth step, expression will be done
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Other): This group will receive the Oketani massage.
  Interventions: Other: Oketani massage group
- Control group (No Intervention): Primipara women in the control group who meet the inclusion criteria will be informed about the study and their consent will be obtained. This group will receive postpartum routine breast care according to health care facility policy. and they will be assessed according to outcome measures in the study

INTERVENTIONS:
Other: Oketani massage group — primipara who meet inclusion criteria and who are assigned to the intervention group will be informed about the study and their consent will be obtained.. Primipara mothers in the intervention group will receive Oketani massage after delivery to enhance successful breastfeeding. The massage is performed using 8 specific hand steps (7 steps for separating the mammary glands and 1 step for expression). Each session lasts 15-20 minutes and is repeated according to the study protocol. the researcher will train primipara relatives to apply Oketani massage after discharge to primipara after discharge. The massage aims to increase milk flow, reduce breast engorgement, improve breast softness, enhance nipple elasticity, and increase maternal comfort and breastfeeding self-efficacy.
  Arms: Intervention group

SUMMARY:
Breastfeeding is essential for infant survival and maternal health; however, many primipara women experience breastfeeding difficulties in the early postpartum period, particularly breast engorgement, ineffective milk transfer, and low breastfeeding self-efficacy, which may compromise successful breastfeeding. Oketani massage is a non-pharmacological, cost-effective breast massage technique developed to enhance milk flow, reduce breast engorgement, and improve maternal comfort during breastfeeding.

This study aims to evaluate the effect of Oketani massage on successful breastfeeding among primipara women. Successful breastfeeding will be assessed through indicators of effective milk transfer, breastfeeding frequency, breast softness after feeding, engorgement prevention and maternal breastfeeding self-efficacy. The findings of this study may support the use of Oketani massage as a supportive nursing intervention to promote successful breastfeeding outcomes in the early postpartum period

ELIGIBILITY:
inclusion criteria:

1. Age between 18 and 35 years
2. Singleton pregnancy
3. Term gestation (>37-40 weeks).
4. Women willing to breast feed
5. The woman will deliver by cesarean section and has relative with her
6. Absence of maternal physical and/ or mental illness that prevents breastfeeding.

The exclusion criteria include:

1. Women with breast problems such as breast tumors, breast surgery and nipple problems
2. Women have obstetric complications as postpartum hemorrhage.
3. Neonatal problems

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The LATCH Assessment sheet | baseline; 2nd time after the 1st six hours after birth and the third time on 1 day of discharge
  It will be adopted from (Jensen et al, 1994) to assess primipara women's need for breastfeeding support, it is numbered from zero to ten, and getting a score of less than ten offers the women's need for more support during breastfeeding. The letters of the acronym LATCH appoint separate areas of assessment: L (Latch) for how well the infant latches onto the breast; A (Audible swallowing) refers the amount of audible swallowing noted while nursing the neonate; T (Type of nipple) for the women's nipple type; C (Comfort) for the women's level of comfort regarding the breast and nipple; and H (Hold) indicates to whether or not the women need help in positioning the infant.
  Scoring system:
  The system assigns a numerical score, 0, 1, or 2, to five key statements. LATCH score of poor (0 to 3), moderate (4 to 7), and good (8 to 10)

SECONDARY OUTCOMES:
Infant Breastfeeding Assessment Tool (IBFAT). | baseline; 2nd time after the 1st six hours after birth and the third time on 1 day of discharge
  It will be adopted from (Matthews, 1988) to assess the infant state and contains four statements as the following: (1) infant readiness to feed/reusability, (2) rooting, (3) fixing (the time needed to latch to the breast), and (4) the sucking pattern.
  Scoring system:
  Each item is scored on a scale of 0-3, with minimum and maximum scores of 0 to 12, respectively. A score of 10-12 refers to completely successful breastfeeding behavior, a score of 7-9 indicates relatively successful breastfeeding behavior and a score of 0-6 suggests unsuccessful breastfeeding behavior.

OTHER OUTCOMES:
The Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF). | baseline; 2nd time after the 1st six hours after birth and the third time after one week
  It will be adopted by (Dennis et al., 2011) to measure breastfeeding confidence. The short form scale contains 14 statements as (I think I can always breastfeed my baby without using formula as a supplement, I think I can always keep wanting to breastfeed, ….. etc) that are scored on a 5-point Likert scale ranging from very confident (score 5) to never confident (score 1). The minimum on this scale is 14 and the maximum possible score is 70. The total scores breastfeeding self-efficacy ranged from 14 to 70 then the level of self-efficacy categorized as the following:
  O Low self-efficacy < 60% (14- 41) O Medium self-efficacy 60% to <75% (42 - 51) O High self-efficacy ≥ 75% (52 - 70).
Six-point engorgement scale | One week post delivery
  It will be adopted from (Hill and Humenick,1994). Breast engorgement was graded on a scale of 1 to 6. Each score represented the following description: (1) soft and no changes in the breast, (2) small changes in the breast, (3) firm and no tender breast, (4) firm and beginning tenderness in the breast, (5) firm and tender of the breast, and (6) very firm and tender.
  Scoring system:
  Score 1 signifies normal breast (no engorgement). Score 2 and 3 signifies mild breast engorgement. Score 4 and 5 signifies moderate breast engorgement. Score 6 signifies severe breast engorgement.

CONTACTS AND LOCATIONS:
Overall Officials: Nasr, Principal Investigator — Faculty of Nursing, Dakahlia Governorate, Mansoura University, Mansoura City, Egypt.
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided